CLINICAL TRIAL: NCT02335281
Title: Efficacy, Durability and Safety of Standardized Fecal Microbiota Transplantation for Severe Inflammatory Bowel Disease
Brief Title: Standardized Fecal Microbiota Transplantation for Inflammatory Bowel Disease
Acronym: SFMT-IBD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yanling Wei (Other)
Responsible Party: Sponsor-Investigator, Yanling Wei, Department of Gastroenterology, Research Institute of Surgery, Da ping Hospital, The Third Military Medical University, Third Military Medical University
Organization: Third Military Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMMU-DP-GI-FMT-001
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Inflammatory Bowel Disease; Ulcerative Colitis; Crohn's Disease
Keywords: Standardized Fecal Microbiota Transplantation; Inflammatory Bowel Disease; Ulcerative Colitis; Crohn's Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standardized FMT (Experimental): The group include 20 patients. They will receive standardized FMT. The FMT was given to mid-gut by nose-jejunum nutrition tube. It was given only once.
  Interventions: Procedure: FMT
- Mesalazine (Active Comparator): This group include 20 patients . The patients will receive traditional medicine of mesalazine treatment.
  Interventions: Drug: Mesalazine

INTERVENTIONS:
Procedure: FMT — Standardized FMT once
  Arms: Standardized FMT
Drug: Mesalazine — 2g Po perday
  Other Names: Mesalamine
  Arms: Mesalazine

SUMMARY:
There are many limitations in the current treatments of Inflammatory bowel disease (IBD). Now the investigators realized that the intestinal microecological is closely associated with the development of IBD. So the standardized fecal microbiota transplantation is considered to be simple but effective emerging therapies for the treatment of IBD. In this project the investigators intend to carry out a single-center, randomized, single-blind clinical intervention study. The investigators will recruit 40 patients with IBD (20 cases of Ulcerative Colitis and 20 cases of Crohn's disease) in China. The patients will be randomly divided into 2 groups, one group will be given treatment of standardized fecal microbiota transplantation, the other will be simply treated with mesalazine, followed up for at least 1 year. The investigators propose to determine the efficiency, durability and safety of Standardized Fecal Microbiota Transplantation for IBD treatment.

DETAILED DESCRIPTION:
In this projects the investigators aim to re-establish a gut balance of intestinal microecological through Standardized Fecal Microbiota Transplantation for IBD (UC and CD). We will establish a standardized isolation, store, and transportion steps of fecal bacteria from donated fresh stool in the laboratory. Then the bacteria will be transplanted to mid-gut by nose-jejunum nutrition tube. Patients in this study will be assigned to receive standardized FMT only once or traditional medicine of mesalazine and would be followed up for at least 1 year. The clinical symptoms, sign, blood tests, abdominal CT, endoscopy and questionnaire will be used to assess the efficiency, durability and safety of Standardized FMT at the start and end of the projects.

ELIGIBILITY:
Inclusion Criteria:

* Severe IBD define as HBI score ≥ 9.
* Moderate IBD define as 7<HBI <9
* Montreal classification: Age > 14 years old, Location L1-3, Behavior B1-3.

Exclusion Criteria:

* Diarrhea activity scores < 3
* Severely active disease with perianal diseases
* Severely active disease with indication of surgery.
* Diagnosis as IBD first time or first year.
* No history of using 5-ASA, biological (antibody), immunomodulatory therapy, corticosteroid therapy

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Clinical remission (defined as HBI score ≦ 4) | up to one year
  Clinical remission defined as HBI score ≦ 4. The endpoint of follow-up is the time of clinical recurrence

SECONDARY OUTCOMES:
Hospitalization days | up to one year
  Hospitalization days from administration to discharge when at clinical remission.

CONTACTS AND LOCATIONS:
Overall Officials: Dongfeng Chen, doctor, Study Director — Third Military Medical University
Locations (1):
- Department of Gastroenterology, Research Institute of Surgery, Da ping Hospital, The Third Military Medical University, Chongqing, Chongqing Municipality, China